CLINICAL TRIAL: NCT02562690
Title: Assessment of Thrombotic Status in Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Hertfordshire (Other)
Collaborators: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Principal Investigator, Diana A Gorog, Professor, University of Hertfordshire
Other Study IDs: RD2014-134
Record Dates: First submitted 2015-09-27; First posted 2015-09-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Coronary Artery Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Coronary Thrombosis
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Coronary Thrombosis | interventions — Thrombelastography; Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Coronary Syndrome: Patients with acute chest pain and persistent ST-segment elevation or new left bundle branch block on the 12 lead ECG. This is termed ST-segment Elevation Myocardial Infarction (STEMI).
  Patients with acute chest pain but without persistent ST-segment elevation. These patients, based on the measurement of cardiac biomarker values (troponin), will be further classified as Non-ST-segment Elevation Myocardial Infarction (NSTEMI) or unstable angina.
  Where possible, all patients will have tests of thrombotic status including thrombin generation assays, TEG and GTT.
  Interventions: Other: Thrombin generation assays, TEG and GTT

INTERVENTIONS:
Other: Thrombin generation assays, TEG and GTT — Thrombin generation assays, Thromboelastography (TEG), and Global Thrombosis Test (GTT)

SUMMARY:
Impaired thrombotic status is associated with adverse cardiovascular events. Patients with acute coronary syndrome (ACS) are at increased cardiovascular risk. The aim of the study is to determine the usefulness of thrombotic status assessment in a large cohort of ACS patients, managed with contemporary treatments, to identify patients at risk of thrombosis and those at risk of bleeding complications.

DETAILED DESCRIPTION:
Patients presenting with acute coronary syndrome (ACS) are at increased risk of future cardiovascular events, despite optimal medical treatment and coronary intervention. Such events are usually caused by increased stickiness of the blood causing a blood clot (thrombus) to block arterial blood vessels in the heart. Much of the medication to prevent recurrent thrombotic events increases the risk of bleeding complications. Identification of patients at recurrent thrombotic risk could allow targeted treatment with potent antithrombotic medications, with less potent agents in others to reduce bleeding. The investigators will assess the stickiness of the blood (i.e. thrombotic status) in patients who are admitted to hospital with ACS; at baseline, at discharge from hospital and at 30 days post hospitalisation. Blood stickiness will be tested using a number of tests of thrombotic status including thrombin generation assays, Thromboelastography (TEG) and the near-patient, point-of-care Global Thrombosis Test (GTT). The results will be evaluated to assess the effect of disease process and clinical state on blood stickiness to gain further understanding of the condition and form the basis for future studies aimed at identifying patients who are at high risk of future cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or over.
2. Patients diagnosed with ACS and free of exclusion criteria below.
3. The patient is willing and able to understand the Patient Information Sheet and provide written informed consent.
4. The patient must agree to comply with the drawing of blood samples for the assessments.

Exclusion Criteria:

1. The patient has, in the opinion of the investigator, significant neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, haemorrhagic, metabolic or other disease likely to confound the study requirements or analyses.
2. The patient has a history of substance abuse or demonstrates signs or clinical features of active substance abuse or psychiatric disease.
3. Alcohol consumption above recommended safe levels (i.e. more than 21 units per week for males, or more than 14 units per week for females) due to the potential effects of high alcohol levels on platelet reactivity.
4. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study.
5. Any major bleeding diathesis or blood dyscrasia (platelets < 70 x 109/l, Hb < 8 g/dl, INR > 1.4, APTT > x 2 UNL, leucocyte count < 3.5 x 109/l, neutrophil count < 1 x 109/l).
6. Currently enrolled in an investigational device or drug trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Coronary Syndrome (ACS) Patients. ACS patients will comprise of patients admitted to hospital with suspected cardiac chest pain and at least 2 of the following 3 criteria of (1) chest pain, (2) ischaemic ECG changes (3) a cardiac troponin measurement exceeding the 99th percentile of a normal reference population (upper reference limit).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Co-primary endpoints of Major Adverse Cardiovascular Events (MACE) and major bleeding | 12 months

SECONDARY OUTCOMES:
Target Lesion Revascularization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Diana A Gorog, MD, PhD, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (1):
- Hertfordshire Cardiology Centre, East and North Hertfordshire NHS Trust, Hertfordshire, United Kingdom

REFERENCES:
- [Derived] Kraler S, Liberale L, Tirandi A, Moriero M, Wang Y, Farag M, Carbone F, Bertolotto MB, Pusterla V, Ramoni D, Ministrini S, Puspitasari YM, Bruno F, Raber L, Di Vece D, Templin C, Muller O, Mach F, Crea F, Camici GG, Lapikova-Bryhinska T, Akhmedov A, von Eckardstein A, Gorog DA, Montecucco F, Luscher TF. The junctional protein associated with coronary artery disease predicts adverse cardiovascular events in patients with acute coronary syndromes at high residual risk. Eur Heart J. 2025 Dec 23:ehaf979. doi: 10.1093/eurheartj/ehaf979. Online ahead of print. PMID 41430589
- [Derived] Farag M, Spinthakis N, Gue YX, Srinivasan M, Sullivan K, Wellsted D, Gorog DA. Impaired endogenous fibrinolysis in ST-segment elevation myocardial infarction patients undergoing primary percutaneous coronary intervention is a predictor of recurrent cardiovascular events: the RISK PPCI study. Eur Heart J. 2019 Jan 14;40(3):295-305. doi: 10.1093/eurheartj/ehy656. PMID 30380032
- [Derived] Farag M, Spinthakis N, Srinivasan M, Sullivan K, Wellsted D, Gorog DA. Morphine Analgesia Pre-PPCI Is Associated with Prothrombotic State, Reduced Spontaneous Reperfusion and Greater Infarct Size. Thromb Haemost. 2018 Mar;118(3):601-612. doi: 10.1055/s-0038-1629896. Epub 2018 Feb 14. PMID 29444530